CLINICAL TRIAL: NCT00036621
Title: A Randomized, Placebo-Controlled Trial of BMS-275291 Given Daily for 12 Months to Women With Stage 1c-IIIA Breast Cancer Receiving Adjuvant Chemotherapy and/or Hormonal Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: CA161-006
Record Dates: First submitted 2002-05-11; First posted 2002-05-13 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-((2S)-2-mercapto-1-oxo-4-(3,4,4- trimethyl-2,5-dioxo-1-imidazolidinyl)butyl)-L-leucyl-N,3- dimethyl-L-Valinamide

INTERVENTIONS:
Drug: BMS-275291

SUMMARY:
This clinical trial will assess whether BMS-275291 can be administered safely in combination with standard adjuvant therapy for early breast cancer and whether plasma concentrations at trough exceed a target minimum.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed pathologic stage 1c-IIIA adenocarcinoma of the breast which has been completely resected.
2. Systemic therapy is planned according to one of the following three regimens:

   * Tamoxifen (20mg) given orally once per day
   * Adriamycin (60 mg/m2 IV on Day 1) plus cyclophosphamide (600mg/m2 IV on Day 1), repeated every 21 days for four courses (to begin within 8 weeks after definitive surgery)
   * Adriamycin (60mg/m2 IV on Day 1) plus cyclophosphamide (600mg/m2 IV on Day 1), repeated every 21 days for four courses, followed by Taxol (175mg/m2 IV on Day 85) repeated every 21 days for four courses (to begin within 8 weeks after definitive surgery).
3. ECOG performance status 0 or 1.
4. Adequate organ function as evidenced by:

   * ANC > 1500/mm3
   * Platelets > 100,000/mm3
   * Serum Creatine < 1.5 ULN
   * Total bilirubin < 1.5 x ULN
   * AST < 2 x ULN
5. Patients to receive adriamycin must have LVEF > 50% or acceptable function per the institutional practice as assessed by MUGA.
6. Signed informed consent.
7. Women age =/> 18 years
8. Patients must have recovered from reversible adverse events of prior surgery and any radiation therapy.
9. Women of childbearing potential must have a serum or urine pregnancy test within 72 hours prior to the start of study medication.

Exclusion Criteria:

1. Patients in whom breast cancer is present at the margin or surgical resection are not eligible in this study. Patients suspicious for residual disease following resection are not eligible.
2. Prior chemotherapy or immunotherapy for breast cancer.
3. Documented metastatic breast cancer.
4. Other malignancy (except carcinoma in situ of the cervix or surgically treated non-melanoma skin cancer) within 5 years of study entry.
5. Pregnant or breastfeeding females.
6. Women of child bearing potential not employing adequate contraception.
7. History of autoimmune diseases such as systemic lupus, rheumatoid arthritis, scleroderma.
8. Any serious underlying medical conditions which would impair the ability ot the patient to receive the planned treatment or which may interfere with the completion of this trial.
9. Planned chemotherapy, hormonal therapy or biological therapy other than those described above. Patients should not be enrolled in any other clinical trials. Use of other investigational agents is not permitted.
10. Any condition that does not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, The Bronx, New York
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Burlington, Vermont
  - Local Institution, Vancouver, Washington
  - Local Institution, Green Bay, Wisconsin